CLINICAL TRIAL: NCT06990009
Title: The Effect of Physical Exercise on Sleep Quality, Quality of Life and Fatigue in Postpartum Women
Brief Title: The Effect of Physical Exercise After Childbirth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ümran erciyes (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor-Investigator, ümran erciyes, Master of Science, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025/183
Record Dates: First submitted 2025-04-12; First posted 2025-05-25 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-04

CONDITIONS: Postpartum
Keywords: exercise; quality of life; fatigue; sleep; postpartum
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: a randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): In line with the Puerperium and Newborn Care Guide, an exercise implementation protocol will be prepared by obtaining the opinion of a group of 10 experts on the appropriateness of the exercises and when they should be started. In this direction, a brochure and a video will be created for the participants to practice the exercises. A pilot study will be conducted in a group of 10 people on the use of the brochure and video, and the brochure and video will be finalized.
  Participants will be asked to do these exercises for 30 minutes a day, five days a week for eight weeks. A reminder message will be sent to the exercise group by the researchers to remind them of the exercises and provide motivation for eight weeks.
  Interventions: Behavioral: exercise
- control (No Intervention): The control group will not receive any intervention and routine care will continue.

INTERVENTIONS:
Behavioral: exercise — In line with the Puerperium and Newborn Care Guide, an exercise implementation protocol will be prepared by obtaining the opinion of a group of 10 experts on the appropriateness of the exercises and when they should be started. In this direction, a brochure and a video will be created for the participants to practice the exercises. A pilot study will be conducted in a group of 10 people on the use of the brochure and video, and the brochure and video will be finalized. Participants will be asked to do these exercises for 30 minutes a day, five days a week for eight weeks. A reminder message will be sent to the exercise group by the researchers to remind them of the exercises and provide motivation for eight weeks.
  Arms: exercise

SUMMARY:
Postpartum women are recommended to engage in physical activity including moderate intensity aerobic and strengthening exercises for at least 150 minutes within one week. The benefits of postpartum exercise include strengthening abdominal muscles, increasing energy, preventing postpartum depression, reducing stress, improving sleep quality and losing excess weight gained during pregnancy. However, activity levels of women who have given birth are reported to be very low, despite the great benefits of exercise on physical and mental health. In a meta-analysis, it was stated that exercise can be used for counseling and therapeutic purposes to improve postpartum quality of life and reduce fatigue.

DETAILED DESCRIPTION:
Although studies evaluating sleep quality, quality of life and fatigue of postpartum women have been found in the literature, no study evaluating the effect of postpartum physical exercise in Turkey has been found yet. Accordingly, this study was planned to evaluate the effect of physical exercise on sleep quality, quality of life and fatigue in postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age
* Be able to read and write in Turkish
* Be in the 24th postpartum hour
* Have had a vaginal delivery
* Have had a single live birth -Have had a single live birth
* Be primiparous
* Have given birth at term -Have given birth at term
* Accept to participate in the study
* Have no musculoskeletal disorder preventing exercise
* Have no chronic disorder preventing exercise
* Using a smart phone

Exclusion Criteria:

* Having a regular exercise program
* Having a baby in intensive care
* Having a psychiatric treatment in the postpartum period
* Being multiparous
* Willing to voluntarily leave the study
* Did not perform the exercises more than two days in a week

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — It is planned in women because it is planned in people who have given birth
Enrollment: 108 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Physical exercise increases sleep quality in postpartum women | 8 week
  Physical exercise improves sleep quality in postpartum women. Participants will be asked to do these exercises for 30 minutes a day, five days a week and for eight weeks in accordance with the brochure and video prepared for the exercise. An evaluation will be made with Pittsburg Sleep Quality Index at the 24th hour and in the fourth week after birth. The final evaluation will be made at the end of the eighth week.
  Pittsburg Sleep Quality Index was developed by Buysse et al. in 1989. Turkish validity and reliability study was conducted by Ağargün et al. in 1996. It consists of a total of 24 questions, 19 of which are answered by the individual and five of which are answered by the relative/roommate. The 19 questions answered by the individual are included in the scoring. It consists of seven components that assess sleep duration, subjective sleep quality, sleep efficiency, sleep latency, the degree to which sleep interferes with daytime activities and the use of sleeping pills.
Physical exercise increases the quality of life in postpartum women | 8 week
  The WHOQOL-BREF-TR will be evaluated at 24 hours and 4 weeks after delivery. The final evaluation will be made at the end of the 8th week. The effect of exercise on quality of life will be evaluated.
  WHOQOL-BREF-TR is a scale developed by the World Health Organization's Quality of Life Group to assess how people perceive their quality of life. The Turkish validity and reliability study of the questionnaire was conducted by Eser and colleagues in 1999. It is a shortened version of the 100-question quality of life scale reduced to 26 questions. The 27th question is a national question. While answering the questions, people are asked to think about the last 15 days of their lives. It is a five-point Likert-type scale. Scores are calculated in four domains and the first two questions are general health assessments and are not used to calculate quality of life.
Physical exercise reduces fatigue in postpartum women | 8 week
  Participants will be asked to do the exercises for 30 minutes a day, five days a week, and for eight weeks. The Piper Fatigue Scale will be used to evaluate the 24th hour and fourth week after birth. The final evaluation will be made at the end of the eighth week. The effect of exercise on reducing fatigue will be evaluated.
  Piper Fatigue Scale: In 1998, it was developed by F. Piper and colleagues. Turkish validity and reliability study was conducted by Can et al. in 2001. It consists of 22 items and four sub-dimensions. When calculating the score, each item is scored between 0-10 and the total score is divided by the number of items. To calculate the subscale scores, the items in each subscale are summed and divided by the number of items in the relevant subscale. A high score on the scale indicates a high level of fatigue. While the total cronbach alpha coefficient of the scale is 0.94, the value of the subscales varies between 0.87-0.91.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay YILMAZ, Study Director — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No